CLINICAL TRIAL: NCT01820871
Title: A Pilot Study of Self Management Using Application for Chronic Disease Care in Real siTuation (SMART) - DM
Brief Title: Self-Management Using Smartphone Application for Type2 DM in Real siTuation (SMART-DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Jongha Park, Study principal investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-DM
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM; smartphone application; serum fasting glucose; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- application arm (Experimental): The patients of application arm have the smartphone application (android) for management of type 2 DM.
  The application contains action plans and alarm system for each situation of serum fasting glucose, blood pressure, body weight, exercise amount, calori intake, medication, etc.
  Interventions: Other: Self-Management Using Smartphone Application for Type2 DM
- conventional arm (Active Comparator): The patients of conventional arm have the booklet for management of type 2 DM. The application contains general medical guideline and knowledge for management of type 2 DM such as,exercise amount, calori intake, medication, etc.
  Interventions: Other: self-management using booklet for management type 2 DM

INTERVENTIONS:
Other: Self-Management Using Smartphone Application for Type2 DM
  Arms: application arm
Other: self-management using booklet for management type 2 DM
  Arms: conventional arm

SUMMARY:
The purpose of this study is to evaluate the effectiveness of smartphone application for management of type 2 diabetes mellitus (DM).

Type 2 DM is an almost incurable chronic disease and continuous management is important for long-term prognosis. However, patient's compliance to conventional medical intervention is generally unsatisfactory and many patients feel difficult to access to the detail medical advice for type 2 DM.

Thus, the investigators developed a smartphone application for giving programed medical intervention to patients according to patients data; blood pressure, fasting blood sugar, body weight, calorie intake,exercise amount, etc.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM using oral hypoglycemic agent
* 6.5% < HbA1c < 10%
* systolic blood pressure > 130 mmHg or diastolic blood pressure > 80 mmHg
* BMI over 23.0
* 20 < age < 70
* smartphone user (android OS based)

Exclusion Criteria:

* Serum fasting glucose > 250 mg/L or post prandial 2 hour serum glucose > 350 mg/L
* systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg
* Diabetes mellitus patient using insulin
* severe chronic diabetic complications (diabetic foot ulcer, severe diabetic retinopathy, diabetic nephropathy with severe proteinuria)
* congestive heart failure (NYHA III-IV or left ventricular ejection fraction < 30%)
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) over 3 times of upper normal limit
* Serum creatinine > 1.5 mg/dL
* refusal to participate in the study
* drug addiction or alcohol addiction
* major psychiatric illness
* steroid treatment or hormonal treatment with changing the drug or drug dosage in 1 month
* changing dosage of antihypertensive agent, oral hypoglycemic agent or lipid lowering agent in 1 month
* malignant cancer
* pregnancy

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
fasting serum glucose and HbA1c | 3months after enrollemnt (day 0-day 90)
  we will check the fasting serum glucose and HbA1C at the day of enrollment (day0)and those at 3months after enrollment (day 90)

SECONDARY OUTCOMES:
body weight and BMI | 3months after enrollemnt (day 0-day 90)
  we will check body weight and BMI at the day of enrollment (day0)and those at 3months after enrollment (day 90)
Lipid profile | 3months after enrollment (day 0-90)
  we will check the lipid profile (total cholesterol, Triglyceride, LDL/HDL cholesterol)at the day of enrollment (day0)and those at 3months after enrollment (day 90)

CONTACTS AND LOCATIONS:
Overall Officials: Jongha Park, MD, Principal Investigator — Inje University
Locations (1):
- Haeundae Paik Hospital, Busan, South Korea